CLINICAL TRIAL: NCT07147816
Title: Effects of Transcutaneous Cervical Spinal Cord Stimulation on Upper Limb Motor Function After Traumatic Brain Injury
Brief Title: Cervical Transcutaneous SCS for TBI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated due to administrative and logistical constraints following the Principal Investigator's transfer to another institution.
Sponsor: Roberto de Freitas (Other)
Collaborators: Chuck Noll Foundation (Unknown)
Responsible Party: Sponsor-Investigator, Roberto de Freitas, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY25060159
Record Dates: First submitted 2025-08-20; First posted 2025-08-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-09

CONDITIONS: Traumatic Brain Injury; TBI (Traumatic Brain Injury)
Keywords: Spinal Cord Stimulation; Transcutaneous Spinal Cord Stimulation; SCS; tSCS
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Prospective, non-randomized, open-label, descriptive, experimental study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Transcutaneous electrical stimulation of the cervical spinal cord (tSCS) (Experimental)
  Interventions: Device: Transcutaneous electrical stimulation of the cervical spinal cord (tSCS)

INTERVENTIONS:
Device: Transcutaneous electrical stimulation of the cervical spinal cord (tSCS) — All participants enrolled in this group will receive non-invasive transcutaneous electrical stimulation of the cervical spinal cord (tSCS) while performing strength, spasticity and motor control assessment tasks. Researchers will assess the immediate effects of tSCS (within the same experimental session) on arm and hand movements in individuals with motor impairments caused by traumatic brain injury.

SUMMARY:
The goal of this study is to test the effects of non-invasive electrical stimulation of the spinal cord (called transcutaneous spinal cord stimulation, or tSCS) on arm and hand movement in people with motor impairments after a traumatic brain injury (TBI). Specifically, tSCS will be delivered using adhesive electrode pads placed on the skin over the upper back. The research team will measure how tSCS affects strength, movement control and muscle spasticity using different tests. Results of this study will help develop future treatments using an implanted (invasive) form of spinal cord stimulation to improve arm and hand function, helping people with TBI become more independent and improve their quality of life.

DETAILED DESCRIPTION:
The main goal of this study is to assess the immediate effects of cervical transcutaneous spinal cord stimulation (tSCS) on arm and hand motor functions after traumatic brain injury (TBI). Specifically, the investigators will assess the immediate effects of tSCS across four different axes: arm and hand strength, arm motor control, joint synergies and spasticity.

The study hypothesis is that tSCS can immediately facilitate voluntary motor output of upper limb muscles by modulating residual descending drive to spinal motoneurons in TBI individuals. In this approach, tSCS targets large-diameter sensory fibers projecting onto motor neuron pools of upper limb muscles. Thus, by modulating the activity of these sensory fibers, the investigators hypothesize that tSCS can immediately increase the excitability of motoneurons receiving residual supraspinal input during movement execution.

Upon completion of this study, the investigators expect to build foundational evidence supporting the use of invasive (e.g. epidural spinal cord stimulation) and non-invasive SCS (tSCS) to improve upper limb motor function in individuals affected by chronic motor impairments after TBI. These results will lay the groundwork for future studies aimed at developing SCS neuroprosthetic devices.

ELIGIBILITY:
Inclusion Criteria:

TRAUMATIC BRAIN INJURY (TBI) SUBJECTS:

* Participants must have a suffered a traumatic brain injury resulting in impairments in arm and hand motor function at least one year prior to enrollment.
* Participants must be between the ages of 21 and 70 years old.

HEALTHY CONTROL SUBJECTS:

* Participants must have full range of motion in their upper limbs;
* Participants must be between the ages of 21 and 70 years old.

Exclusion Criteria:

TRAUMATIC BRAIN INJURY (TBI) SUBJECTS:

* Participants with severe behavioral or cognitive impairments (e.g., aphasia, apraxia, visual neglect) that could preclude their ability to participate in the study.
* Participants diagnosed with Paroxysmal Sympathetic Hyperactivity (PSH);
* Participants with post-TBI heterotopic ossification or tendon contractures that restricts passive range of motion of upper limb joints;
* Participants with uncontrolled epilepsy or untreated seizure disorders;
* Participants with implanted electronic devices, such as pacemakers and spinal cord stimulators;
* Participants taking benzodiazepine for spasticity;
* Participants with serious disease or disorder (ex. neurological condition other than TBI, cancer, severe cardiac or respiratory disease, renal failure, etc.) that could affect their ability to participate in this study.
* Female participants must not be pregnant or breast feeding.
* Evaluation to sign consent form score <12.

HEALTHY CONTROL SUBJECTS:

- Participants who have any serious disease or disorder (e.g. cancer, severe cardiac or respiratory disease, neurological conditions, etc.) or cognitive impairments that could affect their ability to participate in this study.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2025-11-26 (Actual); Primary Completion 2026-01-29 (Actual); Study Completion 2026-01-29 (Actual)

PRIMARY OUTCOMES:
Strength | Immediate (tSCS ON vs tSCS OFF condition within the same experimental session)
  Isometric maximum voluntary contraction (MVC) force of shoulder flexion, shoulder extension, elbow flexion, elbow extension, and hand grip under transcutaneous spinal cord stimulation ON and OFF conditions. MVC force will be compared across transcutaneous spinal cord stimulation ON and OFF conditions within the same experimental session.

SECONDARY OUTCOMES:
Spasticity | Immediate (tSCS ON vs tSCS OFF condition within the same experimental session)
  Spasticity will be measured using the Modified Ashworth Scale (MAS) for the following muscle groups under transcutaneous spinal cord stimulation ON and OFF conditions: shoulder flexors, shoulder extensors, shoulder abductors, shoulder adductors, elbow flexors, elbow extensors, wrist pronators, wrist supinators, wrist flexors, wrist extensors, and finger flexors/extensors. The MAS is a 0-4 ordinal scale that quantifies resistance to passive stretch as a measure of spasticity, with lower scores indicating minimal spasticity and higher scores indicating marked spasticity. The MAS scores will be summed across all muscle groups to create an overall metric quantifying spasticity. MAS scores will be compared across transcutaneous spinal cord stimulation ON and OFF conditions within the same experimental session.
Movement smoothness | Immediate (tSCS ON vs tSCS OFF condition within the same experimental session)
  An exoskeleton robot (KINARM) will be used to assess arm movement smoothness during two-dimensional (2D) reaching tasks under transcutaneous spinal cord stimulation ON and OFF conditions. Movement smoothness will be quantified using log-dimensionless jerk of the hand velocity. Log-dimensionless jerk will be compared across transcutaneous spinal cord stimulation ON and OFF conditions within the same experimental session.
Joint velocity | Immediate (tSCS ON vs tSCS OFF condition within the same experimental session)
  An exoskeleton robot (KINARM) will be used to assess arm joint velocity during two-dimensional (2D) reaching tasks under transcutaneous spinal cord stimulation ON and OFF conditions. Arm joint velocity will be quantified as the ratio between the time required to move the arm from an initial position to a final target and the distance between the positions (m/s). Arm joint velocity will be compared across transcutaneous spinal cord stimulation ON and OFF conditions within the same experimental session.
Discomfort/Pain | Immediate (while tSCS is ON)
  Discomfort and/or pain experienced by participants during transcutaneous spinal cord stimulation will be assessed using a self-reported 0-10 scale, where low values indicate low discomfort/pain, and high values indicate high discomfort/pain.
Join Synergies | Immediate (tSCS ON vs tSCS OFF condition within the same experimental session)
  The "movement combining synergies" and "movement out-of-synergies" subcomponents of the Fugl-Meyer Assessment (FMA) for upper extremity motor function will be used to quantify joint synergies under transcutaneous spinal cord stimulation ON and OFF conditions. The Fugl-Meyer Assessment (FMA) is a performance-based impairment index designed to evaluate upper extremity motor function in individuals with post-stroke hemiparesis. The FMA for upper extremity motor function consists of 33 items, each scored with 0-2 points (0 = cannot perform task, 2 = fully performs task), resulting a maximum score of 66 points . For this study, the subscores from the 'movement combining synergies' and 'movement out-of-synergies' components will be summed to quantify changes in joint synergies. FMA subscores will be compared across transcutaneous spinal cord stimulation ON and OFF conditions within the same experimental session.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto M de Freitas, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared with other researchers for the purpose of data analysis and collaboration.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] de Freitas RM, Sasaki A, Sayenko DG, Masugi Y, Nomura T, Nakazawa K, Milosevic M. Selectivity and excitability of upper-limb muscle activation during cervical transcutaneous spinal cord stimulation in humans. J Appl Physiol (1985). 2021 Aug 1;131(2):746-759. doi: 10.1152/japplphysiol.00132.2021. Epub 2021 Jun 17. PMID 34138648
- [Background] de Freitas RM, Capogrosso M, Nomura T, Milosevic M. Preferential activation of proprioceptive and cutaneous sensory fibers compared to motor fibers during cervical transcutaneous spinal cord stimulation: a computational study. J Neural Eng. 2022 May 17;19(3). doi: 10.1088/1741-2552/ac6a7c. PMID 35472720
- [Background] Inanici F, Brighton LN, Samejima S, Hofstetter CP, Moritz CT. Transcutaneous Spinal Cord Stimulation Restores Hand and Arm Function After Spinal Cord Injury. IEEE Trans Neural Syst Rehabil Eng. 2021;29:310-319. doi: 10.1109/TNSRE.2021.3049133. Epub 2021 Mar 2. PMID 33400652
- [Background] Moritz C, Field-Fote EC, Tefertiller C, van Nes I, Trumbower R, Kalsi-Ryan S, Purcell M, Janssen TWJ, Krassioukov A, Morse LR, Zhao KD, Guest J, Marino RJ, Murray LM, Wecht JM, Rieger M, Pradarelli J, Turner A, D'Amico J, Squair JW, Courtine G. Non-invasive spinal cord electrical stimulation for arm and hand function in chronic tetraplegia: a safety and efficacy trial. Nat Med. 2024 May;30(5):1276-1283. doi: 10.1038/s41591-024-02940-9. Epub 2024 May 20. PMID 38769431
- [Background] Powell MP, Verma N, Sorensen E, Carranza E, Boos A, Fields DP, Roy S, Ensel S, Barra B, Balzer J, Goldsmith J, Friedlander RM, Wittenberg GF, Fisher LE, Krakauer JW, Gerszten PC, Pirondini E, Weber DJ, Capogrosso M. Epidural stimulation of the cervical spinal cord for post-stroke upper-limb paresis. Nat Med. 2023 Mar;29(3):689-699. doi: 10.1038/s41591-022-02202-6. Epub 2023 Feb 20. PMID 36807682